CLINICAL TRIAL: NCT04863300
Title: Evaluation Study of a Collaborative Stepped-Care and Productive Ageing Model for Elderly Mental Wellness in Hong Kong
Brief Title: Collaborative Stepped-Care and Productive Ageing Program for Older People With Depressive Symptoms
Acronym: JCJoyAge2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Aberdeen Kai-fong Welfare Association (Other); Caritas Medical Centre, Hong Kong (Other); Christian Family Service Centre (Other); Haven of Hope Hospital (Other); Hong Kong Christian Service (Other); Hong Kong Sheng Kung Hui Lady MacLehose Centre (Unknown); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Young Women's Christian Association (Other); New Life Psychiatric Rehabilitation Association (Other); St. James' Settlement (Other); The Hong Kong Society for the Aged (Unknown); The Mental Health Association of Hong Kong (Other); Neighbourhood Advice-Action Council (Other); Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EA2003001
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Depressive Symptoms
Keywords: Collaborative stepped care; Peer support; Productive ageing; Early case identification; Indicated prevention; Early treatment; Recovery oriented
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The intervention group will receive a collaborative stepped care programme provided by registered social workers and trained peer supporters from two types of NGOs (aged care or mental health service units) according to level of risks, symptom severity, and intervention response of the clients. Home visits or other format of contact will be delivered by trained peer supporters employed by NGOs to detect and engage hidden cases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in the intervention group will receive a collaborative stepped care programme provided by registered social workers and trained Peer Supporters from aged care service units - the Districts Elderly Community Centres (DECC), and mental health service units - the Integrated Community Centre on Mental Wellness (ICCMW), all are local NGOs. In the collaborative stepped care model (see attachment Table 1), older persons are matched to the intervention module that most suits their current needs. The person does not have to start at the lowest level of intervention to progress to the next level of intervention. Rather, they enter the service with the intervention level aligned to their needs, e.g., level of risks, symptom severity (measured by the Patient Health Questionnaire, PHQ-9), and intervention response. Home visits or other format of contact will be delivered by trained Peer Supporters employed by the NGOs to detect and engage hidden cases.
  Interventions: Behavioral: Collaborative stepped care and peer support

INTERVENTIONS:
Behavioral: Collaborative stepped care and peer support — Case identification will be done through open referral and outreach activities such as street booth, talks, and home visits.
  For older adults with mild depressive symptoms (PHQ-9 score 5-9), 6-8 weeks of indicated prevention with psychoeducation or low-intensity psychotherapy would be provided by the project social workers in DECC. For participants with moderate depressive symptoms (PHQ-9 score 10-14), 6-8 weeks high-intensity clinical intervention, mainly group cognitive behavioral therapy (CBT), would be provided by project social workers from DECC and ICCMW. For those with moderately severe depressive symptoms (PHQ-9 score 15-19), 8-10 weeks individual CBT or group CBT at higher frequency would be provided by the project social workers from ICCMW.
  In the progress review when a client is assessed to meet the discharge criteria, a 2-month exit plan involving a Peer Supporter follow-up is invoked.

SUMMARY:
The Jockey Club Holistic Support Project for Elderly Mental Wellness (JC JoyAge) has developed and implemented a collaborative stepped care model for older persons at-risk of or with depression in four districts in Hong Kong since 2015 (Clinical Trials Identifier: NCT03593889). Results from JC JoyAge show that the collaborative stepped-care model is effective in improving older persons' mental wellness, and the specialised training and engagement of Peer Supporters are effective in building capacity in the community. The proposed impact extension programme lasts for four years (from 2020 to 2023), and the overall goal is to expand the JC JoyAge model to all 18 districts in Hong Kong, to provide integrated and evidence-based mental health services to older adults with subclinical depressive symptoms, with the hope of model adoption in regular service upon project completion.

DETAILED DESCRIPTION:
This four-year extension project includes three main elements: 1) Trainings, including different programmes for social services staff, Mental Wellness Ambassadors, and Peer Supporters; 2) Implementation of JoyAge service model: standardized collaborative stepped-care and Peer Support programmes for prevention and early intervention of depression in older adults; and 3) Public awareness campaign: coordinated programmes to increase mental health literacy and raise public awareness.

Specific goals of the programmes through the above three elements include:

1. To implement JC JoyAge clinical protocol and guidelines to coordinate care among community mental health and aged care services centres for elderly mental wellness in 18 districts;
2. To engage vulnerable and at-risk older adults in the community through productive ageing activities and mental wellbeing self-management training;
3. To enhance the capacity of social service staff in handling elderly depression through specialized and infusion training and knowledge exchange;
4. To raise public awareness and elderly mental health literacy among family members, neighbours, community stakeholders, and the general public to encourage early detection/help-seeking on depressive risk of older adults; and
5. To establish evidence of the effectiveness and cost-effectiveness of JC JoyAge Phase II model.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or above; and
* have depressive symptoms of mild level or above; and
* able to give informed consent to participate

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia; and
* (temporary exclusion criteria) imminent suicidal risk; and
* difficulty in communication

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5239 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depression at 12 months | Baseline and 12-month follow-up
  Depression will be measured by the Patient Health Questionnaire (PHQ-9), a 9-item instrument that incorporates depression diagnostic criteria with other leading major depressive symptoms, and rates the frequency of the symptoms that factor into the scoring severity index. PHQ-9 total score ranges from 0 to 27, higher scores indicate higher levels of depression. Change scores of depression will be calculated by subtract the baseline PHQ-9 score from the follow-up PHQ-9 score, and negative results indicates reduction in depression.
Change from Baseline Anxiety at 12 months | Baseline and 12-month follow-up
  Anxiety will be measured by the Generalized Anxiety Disorder scale (GAD-7), a 7-item scale in which responses to each item are rated on a 4-point Likert scale ranging from 0 to 3. The total score will be used, ranging from 0 to 21. Higher scores indicate higher levels of anxiety symptoms. Change scores of anxiety will be calculated by subtract the baseline GAD-7 score from the follow-up GAD-7 score, and negative results indicates reduction in anxiety.
Change from Baseline Loneliness at 12 months | Baseline and 12-month follow-up
  Loneliness will be measured by the UCLA loneliness scale (UCLA-3), a 3-item self-report scale with each item evaluated with scores ranging from 0 (never) to 3 (often). The total score will be used, ranging from 0 to 9. Higher scores indicate greater loneliness. Change scores of loneliness will be calculated by subtract the baseline UCLA-3 score from the follow-up UCLA-3 score, and negative results indicates reduction in loneliness.
Change from Baseline Self-harm Risk at 12 months | Baseline and 12-month follow-up
  Self-harm risk will be assessed using eight items adapted from the Self-Harm Inventory, providing an overall assessment based on total score and clinical judgement. Social service staff assess participants' risk of self-harm (yes or no answers to 10 items) and harm to others (yes or no answers to 4 items). An overall evaluation of suicidal risk score ranges from 0 (No) to 3 (High). The overall evaluation score will be used. Change scores of self-harm risk will be calculated by subtract the baseline overall risk score from the follow-up risk score, and negative results indicates reduction in self-harm risk.
Change from Baseline Service Usage at 12 months | Baseline and 12-month follow-up
  Client Service Receipt Inventory (CSRI) will be used to collect the current types and level of social services which comprise the care package of each participant, and a locally adapted short version would be developed for this purpose. Participants report frequency of usage of different services in the past month when filling the questionnaire, higher frequency indicates more usage of that particular service.

SECONDARY OUTCOMES:
Change from Baseline Daily Activities at 12 months | Baseline and 12-month follow-up
  A semi-structured interview asking clients about their typical day activities in three domains: physical, social, and mental. A combination of being active in at least two domains would be used as one of the exit criteria. The changes of total numbers of activities reported will be calculated.
Change from Baseline Cognition at 12 months | Baseline and 12-month follow-up
  Cognition will be measured by the Hong Kong Montreal Cognitive Assessment 5-Minute Protocol (HK-MoCA 5-Min). It is a validated and reliable cognitive screen for stroke and transient ischemic attack, brief and highly feasible for telephone administration. It includes four items examining attention, verbal learning and memory, executive functions/language, and orientation extracted from the MoCA. Total scores range between 0 and 30, with higher scores indicating better cognition. Change scores of cognition will be calculated by subtract the baseline HK-MoCA 5-Min score from the follow-up score, and positive results indicates improvements in cognition.
Change from Baseline Social Network at 12 months | Baseline and 12-month follow-up
  Social support network is measured by a self-developed questionnaire asking participants to list out names of people who they would turn to (a) when they feel down, and (b) when they need help for trivial things. Participants can report up to 5 people to each condition. More people they can turn to indicates a wider social support network. Change in social support network will be calculated by subtract the baseline number of persons who they can turn to help from the follow-up number, positive results indicates increase in social support network.
Change from Baseline Health-related Quality of Life at 12 months | Baseline and 12-month follow-up
  Health-related quality of life will be measured by the EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L). The EQ-5D-5L is a generic preference-based measure of health on five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels (5L) of problems. The traditional Chinese version for Hong Kong developed by EuroQol Group will be used. Results will be presented by the EQ-5D-5L index value.
Change from Baseline Self-rated Health at 12 months | Baseline and 12-month follow-up
  A visual analogue scale (EQ VAS) will be used for participants to rate their general health from 0 to 100. Change scores of overall self-rated health will be calculated by subtract the baseline EQ VAS from the follow-up EQ VAS score, and positive results indicates improvement in self-rated health.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Lum, PhD, Principal Investigator — The University of Hong Kong
Locations (43):
- Hong Kong (43):
  - Aberdeen Kaifong Welfare Association Services Centre, Hong Kong
  - Baptist Oi Kwan Social Service Integrated Community Centre for Mental Wellness (Kwai Tsing), Hong Kong
  - Baptist Oi Kwan Social Service, Hong Kong
  - Caritas Cheng Shing Fung District Elderly Centre (Sham Shui Po), Hong Kong
  - Caritas District Elderly Centre - Yuen Long(Tin Chak Centre), Hong Kong
  - Caritas Wellness Link - North District, Hong Kong
  - Caritas Wellness Link Tsuen Wan, Hong Kong
  - Chan Tseng Hsi Kwai Chung District Elderly Community Centre, Hong Kong
  - Christian Family Service Centre (Kwun Tong), Hong Kong
  - Christian Family Service Centre Wellness Zone - Integrated Community Centre for Mental Wellness, Hong Kong
  - Chuk Yuen Canon Martin District Elderly Community Centre_Wai Yuen House, Hong Kong
  - Ellen Li District Elderly Community Centre - Yung Shing Shopping Centre, Hong Kong
  - Fong Shu Chuen District Elderly Community Centre, Hong Kong
  - H.K.S.K.H. Lady MacLehose Centre Dr. Lam Chik Suen District Elderly Community Centre, Hong Kong
  - H.K.S.K.H. Lok Man Alice Kwok Integrated Service Centre, Hong Kong
  - H.K.S.K.H. Western District Elderly Community Centre - Integrated Home Care Services Team, Hong Kong
  - Haven of Hope Christian Service, Hong Kong
  - Hong Kong Christian Service Bliss District Elderly Community Centre, Hong Kong
  - Jockey Club Wong Chi Keung District Elderly Community Centre - Aberdeen, Hong Kong
  - Neighbourhood Advice-action Council (Shan King) Community Nursing Services (CNS) Centre, Hong Kong
  - New Life Psychiatric Rehabilitation Association (Sha Tin), Hong Kong
  - New Life Psychiatric Rehabilitation Association (Tuen Mun), Hong Kong
  - New Life Psychiatric Rehabilitation Association (Yau Tsim Mong), Hong Kong
  - New Life Psychiatric Rehabilitation Association Islands District, Hong Kong
  - New Life Psychiatric Rehabilitation Association The Wellness Centre (Tin Shui Wai), Hong Kong
  - S.K.H. Holy Carpenter Church District Elderly Community Centre (Kowloon), Hong Kong
  - Sage Eastern District Elderly Community Centre, Hong Kong
  - Sage Tsuen Wan District Elderly Community Centre, Hong Kong
  - Shun On District Elderly Community Centre, Hong Kong
  - St. James' Settlement Central & Western District Elderly Community Centre, Hong Kong
  - St. James' Settlement Wan Chai District Elderly Community Centre, Hong Kong
  - The Mental Health Association of Hong Kong Amity Place, Hong Kong
  - The Mental Health Association of Hong Kong Tai Po District, Hong Kong
  - The Neighbourhood Advice-Action Council, Hong Kong
  - The Neighbourhood Advice-Action Counil Tung Chung Intergrated Service Centre, Hong Kong
  - The Salvation Army Tai Po Multi-service Centre for Senior Citizens, Hong Kong
  - The Society of Rehabilitation and Crime Prevention, Hong Kong, Hong Kong
  - The Wellness Centre, New Life Psychiatric Rehabilitation Association (Kwai Chung), Hong Kong
  - Tseung Kwan O Aged Care Complex, Jockey Club District Elderly Community Centre cum Day Care Unit, Hong Kong
  - Tung Wah Group of Hospitals Wilson T.S. Wang District Elderly Community Centre, Hong Kong
  - TWGHs Lok Hong Integrated Community Centre for Mental Wellness, Hong Kong
  - Wong Cho Tong District Elderly Community Centre, Hong Kong
  - YWCA Ming Yue District Elderly Community Centre, Hong Kong

REFERENCES:
- [Derived] Wong SMY, Leung DKY, Liu T, Ng ZLY, Wong GHY, Chan WC, Lum TYS. Comorbid anxiety, loneliness, and chronic pain as predictors of intervention outcomes for subclinical depressive symptoms in older adults: evidence from a large community-based study in Hong Kong. BMC Psychiatry. 2024 Nov 21;24(1):839. doi: 10.1186/s12888-024-06281-2. PMID 39574082

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04863300/Prot_SAP_ICF_000.pdf